CLINICAL TRIAL: NCT04428554
Title: Consolidative Radiotherapy for Metastatic Urothelial Bladder Cancer Patients Without Progression and With no More Than Three Residual Metastatic Lesions Following First Line Systemic Therapy: a Prospective Randomized Comparative Phase II Trial
Brief Title: Consolidative Radiotherapy for Metastatic Urothelial Bladder Cancer Patients Without Progression and With no More Than Three Residual Metastatic Lesions Following First Line Systemic Therapy
Acronym: BLAD-RAD01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19 URO 15
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Urothelial Bladder Cancer
Keywords: Urothelial bladder cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Standard of care
- Experimental arm (Experimental)
  Interventions: Radiation: Experimental arm

INTERVENTIONS:
Radiation: Experimental arm — Consolidative radiotherapy (pelvic irradiation and/or metastases irradiation) + standard of care +/- previous transurethral resection of bladder tumor
  Arms: Experimental arm

SUMMARY:
This is a Phase II, multicenter, randomized open-label and comparative study that has been designed to evaluate whether local consolidative radiotherapy in addition to standard of care improves overall survival as compared with standard of care in patients with regional and/or distant metastatic urothelial bladder cancer who have no disease progression and with no more than three residual distant metastatic lesions following the initial phase of first-line systemic therapy.

Each patient will be followed during 4 years from the date of randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
3. Urothelial bladder cancer histologically proven (both pure urothelial cancers and mixed histologic features are allowed)
4. Metastatic patients to regional nodes (Tx,N1-N3,M0) and/or distant sites (Tx,Nx,M1a-M1b) documented with contrast-enhanced CT-scanner of the chest, abdomen and pelvis, either de novo or presenting first regional/distant relapse following cystectomy (with no local recurrence in the cystectomy bed)
5. Completion of the initial phase (4-6 cycles) of 1st line metastatic treatment (systemic therapy by chemotherapy and/or immunotherapy by immune check-point inhibitor according to standard recommendations). Patients having started maintenance therapy are eligible.
6. No disease progression after the initial phase of first-line metastatic systemic therapy according to RECIST v1.1
7. No more than 3 residual distant metastatic lesions following the initial phase of first-line metastatic systemic therapy:

   1. Regional nodes (below aortic bifurcation) are not included in the count of distant metastatic lesions
   2. The number of distant residual lesions is determined on the basis of the imaging modality for tumor response assessment performed after systemic treatment according to local habits (CT-scan or 18FDG PET-CT if performed):

      In case of response assessment by CT-scanner only: residual lesions are all remaining visible lesions In case of response assessment by additional 18FDG PET-CT: residual lesions are only the lesions with residual hyperfixation
   3. Regarding distant lymph nodes metastases:

      * If evaluation is performed by CT-scanner only, residual lymph nodes are considered pathological according to one or several criteria among: Short axis ≥ 1cm/Central necrosis/Heterogeneous contrast enhancement
      * Residual para-aortic nodes involvement accounts for one lesion, even if several para-aortic nodes are involved.
      * Other nodes: each involved node accounts for one lesion.
8. Residual distant metastases (if applicable) eligible for SBRT in terms of dose constraints to the organs at risk, with no prior radiotherapy interfering with SBRT
9. 8 weeks or less between last cycle of the initial phase of systemic treatment and randomization
10. No contraindication to pelvic radiotherapy
11. Signed informed consent
12. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol
13. Patient affiliated to a Social Health Insurance in France

Exclusion Criteria:

1. Non-transitional cell histology (Squamous cell carcinoma, adenocarcinoma or neuroendocrine carcinoma of the bladder)
2. Brain metastases before systemic treatment
3. Liver metastases before systemic treatment
4. Absence of target to be irradiated (i.e. previous cystectomy + no residual distant lesions following systemic treatment + no pelvic or para-aortic nodes at metastatic presentation)
5. Patient with relapse following definitive chemoradiation of the bladder
6. Local recurrence in the cystectomy bed following cystectomy
7. Previous pelvic irradiation
8. Prior radiotherapy near the residual metastatic lesions precluding ablative SBRT
9. Active inflammatory bowel disease
10. Contraindication to SBRT of a lesion due to organ dysfunction; in particular, patients with lung lesions and documented or suspected interstitial lung disease should not be included
11. History of scleroderma
12. Current or past history of second neoplasm diagnosed within the last 5 years (except basocellular carcinoma and prostate cancer incidentally discovered during previous cystoprostatetectomy and pelvic lymph node dissection and with a good prognosis [T stage <pT3b and Gleason <8 and pN- and post-operative PSA <0.1 ng/mL])
13. Pregnancy or breast feeding or inadequate contraceptive measures
14. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
16. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).
17. Concurrent enrolment in another interventional therapeutic clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 4 years for each patient

SECONDARY OUTCOMES:
Progression Free Survival | 4 years for each patient
Safety will be assessed by the toxicity grading of the National Cancer Institute (NCI-CTCAE v5) | 4 years for each patient
Quality of life will be evaluated by the EORTC QLQ-C-30 questionnaire | 4 years for each patient

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Clinique Claude Bernard, Albi
  - Institut de Cancerologie de L'Ouest, Angers
  - CHU Besançon, Besançon
  - Institut Bergonie, Bordeaux
  - CHRU Brest, Brest
  - Clinique Pasteur-Lanroze, Brest
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Andrée Dutreix, Dunkirk
  - Centre Oscar Lambret, Lille
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Institut Curie, Paris
  - Groupement de Radiothérapie et d'Oncologie des Pyrénées, Pau
  - Institut de Cancerologie de L'Ouest, Saint-Herblain
  - HIA Bégin, Saint-Mandé
  - Institut de Cancerologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif